CLINICAL TRIAL: NCT00785629
Title: A Double Blind Randomized Placebo Controlled Trial of Maintenance of Normal Serum Phosphorus in Chronic Kidney Disease (CKD)
Brief Title: A Double Blind Randomized Placebo Trial of Maintenance of Normal Serum Phosphorus in CKD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Denver Nephrologists, P.C. (Other)
Collaborators: Shire (Industry); Fresenius Medical Care North America (Industry); Genzyme, a Sanofi Company (Industry); Novartis Pharmaceuticals (Industry); DaVita, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PNT001
Record Dates: First submitted 2008-11-04; First posted 2008-11-05 (Estimated); Results first posted 2012-10-30 (Estimated); Last update posted 2012-10-30 (Estimated); Status verified 2012-09

CONDITIONS: Chronic Kidney Disease
Keywords: phosphorus; secondary hyperparathyroidism; vascular calcification
MeSH Terms: conditions — Renal Insufficiency, Chronic; Hyperparathyroidism, Secondary; Vascular Calcification | interventions — calcium acetate; lanthanum carbonate; Sevelamer

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Calcium Acetate (Active Comparator): 667 mg with meals
  Interventions: Drug: Calcium acetate
- Lanthanum Carbonate (Active Comparator): 500 mg with meals
  Interventions: Drug: Lanthanum Carbonate
- Sevelamer Carbonate (Active Comparator): 800 mg with meals
  Interventions: Drug: Sevelamer Carbonate
- Placebo (Placebo Comparator): with meals
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Calcium acetate
  Arms: Calcium Acetate
Drug: Lanthanum Carbonate
  Other Names: Fosrenol
  Arms: Lanthanum Carbonate
Drug: Sevelamer Carbonate
  Other Names: Renvela
  Arms: Sevelamer Carbonate
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the ability of 3 commercially available phosphorus binders (calcium acetate, sevelamer carbonate, and lanthanum carbonate) to achieve and maintain a phosphorus level in the normal range in patients with chronic kidney disease.

DETAILED DESCRIPTION:
It is the specific aim of this pilot study to assess the feasibility of achieving and maintaining a serum P less than or equal to 3.5 mg/dL (1.13 mmol/L) in patients with eGFR >20 and <45 mL/min with any of the 3 commercially available P lowering agents (calcium acetate, sevelamer carbonate, or lanthanum carbonate). Results of this study will clarify the degree of separation in serum P that can be achieved with the use of P lowering agents and the current standard of care (P binder initiation when P > 5.5 mg/dL or 1.78 mmol/L). Furthermore, this knowledge, combined with analyses of the secondary aims and outcomes of interest, will serve to facilitate the design of a properly powered, randomized, placebo controlled clinical outcomes trial that will firmly establish the necessity of achieving a specific target P in patients with CKD. The secondary aims of this pilot study are to provide insight into the optimal detection of progression of abnormalities in mineral metabolism and their relationship to vascular disease in CKD. The tertiary aim is to evaluate long term outcomes related to phosphorus normalization with respect to renal replacement therapy or death.

ELIGIBILITY:
Inclusion Criteria:

* Men or women > 18 years of age;
* Has signed and dated the most recent informed consent form approved by an IRB;
* Will, in the opinion of the PI, be compliant with prescribed phosphate binder therapy;
* Must be able to communicate with the investigator, and be able to understand and comply with the requirements of the study;
* Has a life expectancy >12 months;
* An eGFR rate (estimated by the MDRD equation) ≥ 20 and ≤ 45 mL/min/1.73m2 obtained by screening laboratory values and in the opinion of the investigator felt to have CKD without evidence of recent acute kidney injury or unexpected decline in renal function;
* A screening serum phosphorus value > 3.5 mg/dL and ≤ 6.0 mg/dL;
* Must consume a minimum of 2 meals per day and be willing to avoid intentional changes in diet;
* Women of child bearing potential must be practicing an acceptable form of birth control.

Exclusion Criteria:

* Receiving or has received an investigational drug (or is currently using an investigational device) within 30 days prior to baseline;
* Subject is pregnant, is breast feeding or is of child bearing potential and not using acceptable birth control measures;
* Has had a previous renal transplant;
* Has a chronic reliance on enemas or laxatives;
* Has a known sensitivity or previous intolerance to any of the products to be administered during the study;
* Clinical evidence of active malignancy and/or receiving systemic chemotherapy/radiotherapy with the exception of basal cell or squamous carcinoma of the skin;
* Currently has an active infection or is being treated with antibiotics (within 14 days prior to baseline);
* Has been hospitalized within 30 days prior to baseline (with the exception of hospitalizations due to vascular access procedures);
* Any surgical or medical condition which might significantly alter the function of phosphorus binders or which may jeopardize the subject in case of participation in the study. The investigator should be guided by evidence of any of the following: Severe gastrointestinal motility disorder,Bowel obstruction,Dysphagia or other disorders of swallowing, Acute peptic ulcer, Ulcerative colitis or Crohn's disease, History of major gastrointestinal tract surgery, Severe malabsorption;
* Currently taking any of the following within 14 days prior to baseline; Calcitriol or its analogs, Cinacalcet hydrochloride, Medications prescribed for the purpose of phosphorus binding;
* Screening serum intact PTH >500 pg/mL;
* Screening corrected calcium < 8.0 mg/dL or > 10.4 mg/dL;
* Uncontrolled hyperlipidemia in the opinion of the PI;
* Initiation of chronic maintenance hemodialysis planned within 12 months;
* Relocation to another area planned within 12 months;
* Has a known history of immunodeficiency diseases, including a positive HIV test result;
* Active drug or alcohol dependence or abuse (excluding tobacco use) within the 12 months prior to dosing or evidence of such abuse;
* Evidence of active liver disease with AST or ALT levels greater than 3X the upper limit of normal;
* Has had a major cardiovascular event within 180 days of screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2009-02; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Geoffrey A Block, MD, Principal Investigator — Denver Nephrologists, PC
Locations (1):
- Denver Nephrologists, PC, Denver, Colorado, United States

REFERENCES:
- [Derived] Natale P, Green SC, Ruospo M, Craig JC, Vecchio M, Elder GJ, Strippoli GF. Phosphate binders for preventing and treating chronic kidney disease-mineral and bone disorder (CKD-MBD). Cochrane Database Syst Rev. 2025 Jun 27;6(6):CD006023. doi: 10.1002/14651858.CD006023.pub4. PMID 40576086
- [Derived] Dougher CE, Rifkin DE, Anderson CA, Smits G, Persky MS, Block GA, Ix JH. Spot urine sodium measurements do not accurately estimate dietary sodium intake in chronic kidney disease. Am J Clin Nutr. 2016 Aug;104(2):298-305. doi: 10.3945/ajcn.115.127423. Epub 2016 Jun 29. PMID 27357090

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Single center private practice single specialty clinic, Enrollment Feb 2009 thru September 2010
Pre-assignment Details: Consecutive CKD patients with eGFR 20- 45 ml/min with serum Phosphorus >3.5 < 6.0. Stratified by diabetic status. 3 subjects were enrolled but did not receive study medication due to withdrawal prior to starting medication.
Groups:
- Calcium Acetate: phosphate binder : starting dose 667mg;titrations to 2668mg QAC
- Sevelamer Carbonate: phosphate binder : starting dose 800mg; titrations to 3200mg QAC
- Lanthanum Carbonate: phosphate binder : starting dose 500mg; titrations to 1500mg QAC
Period: Overall Study
Arm/Group | Calcium Acetate | Sevelamer Carbonate | Lanthanum Carbonate | Placebo
Started | 30 | 30 | 28 | 57
Completed | 22 (8 not completed) | 25 (5 not completed) | 18 (10 not completed) | 41 (16 not completed)
Not Completed | 8 | 5 | 10 | 16
Not completed — Adverse Event | 2 | 1 | 1 | 5
Not completed — Protocol Violation | 1 | 2 | 4 | 5
Not completed — administrative decision | 5 | 1 | 3 | 4
Not completed — Withdrawal by Subject | 0 | 1 | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Calcium Acetate | Sevelamer Carbonate | Lanthanum Carbonate | Placebo | Total
Number analyzed (Participants) | 30 | 30 | 28 | 57 | 145
Age Continuous [Mean (Standard Deviation); unit: years] | 68 (12) | 66 (12) | 70 (10) | 65 (12) | 67 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 15 | 13 | 29 | 71
  Male | 16 | 15 | 15 | 28 | 74
Region of Enrollment [Number; unit: participants]
  United States | 30 | 30 | 28 | 57 | 145

OUTCOME MEASURES:

1. Primary Outcome: Serum Phosphorus
Description: mean serum phosphorus from months 3-9
Time Frame: months 3-9
Population: ITT analysis was ALL active patients combined versus all placebo patients combined
Measure: Mean (Standard Deviation); unit: mg/dL
Groups:
- All Active Treated Patients: All actively treated patients
- All Placebo Treated Patients: All placebo treated patients
Arm/Group | All Active Treated Patients | All Placebo Treated Patients
Number analyzed (Participants) | 88 | 57
mg/dL | 3.9 (0.4) | 4.2 (0.4)

ADVERSE EVENTS:
Time Frame: Enrollment until 14 days post end of study (last dose)
Arm/Group | Placebo | Lanthanum Carbonate | Sevelamer Carbonate | Calcium Acetate
Serious Adverse Events (participants affected / at risk) | 8/57 | 6/28 | 8/30 | 4/30
Other Adverse Events (participants affected / at risk) | 43/57 | 21/28 | 25/30 | 26/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=57) | Lanthanum Carbonate (N=28) | Sevelamer Carbonate (N=30) | Calcium Acetate (N=30)
Hypothyroidism (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peritoneal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Vascular access complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Transient Ischemic Attack (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Acute Kidney Injury (Renal and urinary disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Pulmonary Edema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thromboembolic Event (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
visceral arterial ischemia (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Total knee replacement (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastric lap banding (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
left ventricular systolic dysfunction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
right ventricular dysfunction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
vitreous hemorrhage (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Other: digitalis toxicity (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
hypergylcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
altered mental status (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
stroke (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=57) | Lanthanum Carbonate (N=28) | Sevelamer Carbonate (N=30) | Calcium Acetate (N=30)
anemia (Blood and lymphatic system disorders) | 4 (4) | 1 (1) | 0 (0) | 2 (2)
conduction disorder (Cardiac disorders) | 1 (1) | 2 (2) | 1 (1) | 1 (1)
left ventricular systolic dysfuction (Cardiac disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
sinus bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
hyperparathyroidism (Endocrine disorders) | 5 (5) | 0 (0) | 4 (4) | 1 (1)
abdominal pain (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0) | 1 (1)
constipation (Gastrointestinal disorders) | 2 (2) | 3 (3) | 7 (7) | 6 (6)
diarrhea (Gastrointestinal disorders) | 6 (6) | 7 (7) | 2 (2) | 3 (3)
dyspepsia (Gastrointestinal disorders) | 3 (3) | 1 (1) | 2 (2) | 3 (3)
enterocolitis (Gastrointestinal disorders) | 4 (4) | 0 (0) | 0 (0) | 1 (1)
flatulence (Gastrointestinal disorders) | 2 (2) | 1 (1) | 3 (3) | 0 (0)
nausea (Gastrointestinal disorders) | 1 (1) | 3 (3) | 3 (3) | 1 (1)
vomiting (Gastrointestinal disorders) | 1 (1) | 6 (6) | 1 (1) | 0 (0)
edema limbs (General disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
pneumonia (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
sinusitis (Infections and infestations) | 4 (4) | 2 (2) | 0 (0) | 0 (0)
soft tissue infections (Infections and infestations) | 3 (3) | 3 (3) | 3 (3) | 0 (0)
upper respiratory infection (Infections and infestations) | 4 (4) | 4 (4) | 2 (2) | 3 (3)
urinary tract infection (Infections and infestations) | 3 (3) | 0 (0) | 3 (3) | 4 (4)
fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 2 (2) | 1 (1)
acidosis (Metabolism and nutrition disorders) | 6 (6) | 3 (3) | 1 (1) | 1 (1)
hypercalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 5 (5)
hyperkalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
hypoglycemia (Metabolism and nutrition disorders) | 5 (5) | 1 (1) | 1 (1) | 0 (0)
arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
arthritis (Musculoskeletal and connective tissue disorders) | 8 (8) | 0 (0) | 4 (4) | 1 (1)
back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
myalgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1) | 1 (1) | 1 (1)
pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
syncope (Nervous system disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
acute kidney injury (Renal and urinary disorders) | 8 (8) | 7 (7) | 4 (4) | 7 (7)
bronchospasm (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1) | 2 (2)
dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
other: laceration (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
pruritis (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
rash- maculo-papular (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)

LIMITATIONS AND CAVEATS:
Single center study; Modest size of study; pilot study not powered to detect differences among subgroups of actively treated patients

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less